CLINICAL TRIAL: NCT01642498
Title: ROX CONTROL HTN Study: A Prospective, Randomized, Open-Label, Multicenter Study to Evaluate the ROX Coupler in Patients With Resistant Hypertension
Brief Title: A Multicenter Study to Evaluate the ROX Arteriovenous Coupler in Patients With Treatment-Resistant Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ROX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RH-02
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Hypertension; Resistant Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): ROX Coupler + continuing standard antihypertensive medications
  Interventions: Device: ROX COUPLER
- Group B (No Intervention): Continuing standard antihypertensive medications

INTERVENTIONS:
Device: ROX COUPLER — The COUPLER will be used to create an arteriovenous fistula in the iliac region (between the iliac artery and vein).
  Arms: Group A

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the ROX COUPLER in patients with treatment-resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of treatment-resistant hypertension must be made on the basis of current findings, medical history, and physical examination

Exclusion Criteria:

* Any serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the study, comply with follow-up requirements or impact the scientific integrity of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mean office SBP | Baseline, 6 months
  Change in mean office SBP at six months as compared to Baseline

SECONDARY OUTCOMES:
Change in mean office DBP | Baseline, 6 months
  Change in mean office DBP at six months as compared to Baseline

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (2):
  - ZNA - Cardio Middleheim, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
- Germany (3):
  - Universitätsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Hypertoniezentrum Marburg, Marburg
- Greece (2):
  - G. Gennimatas General Hospital of Athens, Athens
  - Hippokration General Hospital of Athens, Athens
- Ireland (2):
  - Connolly Hospital, Blanchardstown, Dublin
  - Beaumont Hospital, Dublin
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Poland (2):
  - Jagiellonian University Collegium Medicum, Krakow
  - Institute of Cardiology - Warsaw, Warsaw
- United Kingdom (6):
  - Eastbourne District General Hospital, Eastbourne, England
  - Queen Mary University of London, London, England
  - Royal Bromptom, London, England
  - St. Helier Hospital, Carshalton, Surrey England
  - University Hospital of Wales, Cardiff, Wales
  - University Hospitals of Leicester - Glenfield Hospital, Leicester

REFERENCES:
- [Derived] Lobo MD, Ott C, Sobotka PA, Saxena M, Stanton A, Cockcroft JR, Sulke N, Dolan E, van der Giet M, Hoyer J, Furniss SS, Foran JP, Witkowski A, Januszewicz A, Schoors D, Tsioufis K, Rensing BJ, Scott B, Ng GA, Schmieder RE. Central Iliac Arteriovenous Anastomosis for Uncontrolled Hypertension: One-Year Results From the ROX CONTROL HTN Trial. Hypertension. 2017 Dec;70(6):1099-1105. doi: 10.1161/HYPERTENSIONAHA.117.10142. Epub 2017 Oct 23. PMID 29061728
- [Derived] Ott C, Lobo MD, Sobotka PA, Mahfoud F, Stanton A, Cockcroft J, Sulke N, Dolan E, van der Giet M, Hoyer J, Furniss SS, Foran JP, Witkowski A, Januszewicz A, Schoors D, Tsioufis K, Rensing BJ, Saxena M, Scott B, Ng GA, Achenbach S, Schmieder RE. Effect of Arteriovenous Anastomosis on Blood Pressure Reduction in Patients With Isolated Systolic Hypertension Compared With Combined Hypertension. J Am Heart Assoc. 2016 Dec 21;5(12):e004234. doi: 10.1161/JAHA.116.004234. PMID 28003251
- [Derived] Lobo MD, Sobotka PA, Stanton A, Cockcroft JR, Sulke N, Dolan E, van der Giet M, Hoyer J, Furniss SS, Foran JP, Witkowski A, Januszewicz A, Schoors D, Tsioufis K, Rensing BJ, Scott B, Ng GA, Ott C, Schmieder RE; ROX CONTROL HTN Investigators. Central arteriovenous anastomosis for the treatment of patients with uncontrolled hypertension (the ROX CONTROL HTN study): a randomised controlled trial. Lancet. 2015 Apr 25;385(9978):1634-41. doi: 10.1016/S0140-6736(14)62053-5. Epub 2015 Jan 23. PMID 25620016
- [Derived] Foran JP, Jain AK, Casserly IP, Kandzari DE, Rocha-Singh KJ, Witkowski A, Katzen BT, Deaton D, Balmforth P, Sobotka PA. The ROX coupler: creation of a fixed iliac arteriovenous anastomosis for the treatment of uncontrolled systemic arterial hypertension, exploiting the physical properties of the arterial vasculature. Catheter Cardiovasc Interv. 2015 Apr;85(5):880-6. doi: 10.1002/ccd.25707. Epub 2014 Nov 1. PMID 25345578